CLINICAL TRIAL: NCT01784575
Title: IDEAS for a Healthy Baby: Reducing Disparities in Consumer Use of Publicly Reported Quality Data
Brief Title: Increasing Use of Publicly Reported Pediatric Quality Data
Acronym: IDEAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R21HS021864-01 (AHRQ); R21HS021864-01 (AHRQ)
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Pregnancy
Keywords: Quality of care; Pediatric; Pregnancy; Low-income; Low literacy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Navigator Intervention (Experimental): The Patient Navigator Intervention arm will have two 20 minute interactive sessions with a patient navigator in which they will learn about quality measures and view scores on the Massachusetts Health Quality Partner's website.
  Interventions: Other: Patient Navigator Intervention
- Control (Active Comparator): The control arm will receive an information pamphlet about health care quality.
  Interventions: Other: Patient Navigator Intervention

INTERVENTIONS:
Other: Patient Navigator Intervention — The Patient Navigator Intervention will include 2 - 20 minute sessions with a patient navigator in which women are shown publicly available health care quality data about local pediatric practices on a non-profit quality collaborative's web site.

SUMMARY:
Numerous factors prevent consumers from making effective use of publicly reported information about the quality of health care, including limited recognition that quality of care varies between physicians, lack of awareness of the existing quality websites, limited internet access, and low health literacy and numeracy. In the proposed randomized controlled trial we will evaluate the impact of providing assistance for using and interpreting information about the quality of pediatric care on the Massachusetts Health Quality Partners Quality Insights website among a population of low income pregnant women. Results of the study will advance our understanding of effective strategies for overcoming barriers to using publicly reported information among vulnerable populations.

DETAILED DESCRIPTION:
Efforts to increase transparency regarding health care quality and safety are partially guided by the belief that making performance information publicly available will enable patients to make more informed choices. Although the amount of information reported on websites and through other channels has increased dramatically, use by consumers remains limited and largely restricted to white, college educated and middle aged consumers. There are many barriers that prevent patients from making effective use of current public reporting websites, including failure to recognize that quality may vary between providers, lack of awareness of publicly reported data, limited internet access, and low health literacy and numeracy. Innovative approaches are therefore needed to overcome barriers to using these data, particularly in vulnerable populations, to ensure a health care system in which every consumer can benefit from public reporting. Patient navigators have helped patients take greater advantage of the complex health care delivery environment, and use of patient navigators may be an effective approach to engage consumers and to help them to interpret the information presented in public reports.

The scientific aims of the study are: 1) to test the efficacy of an office-based patient navigator to assist low income pregnant women in using publicly reported data to select a pediatric care provider; 2) to assess the efficacy of the intervention in subgroups defined by parity, race/ethnicity, and health literacy; 3) to evaluate the importance of publicly reported information about quality compared to other factors when selecting a pediatric provider; and 4) to assess the intervention's impact on self-management of health care. English speaking women ages 16-45 attending the prenatal clinic at a large urban medical center will be recruited, enrolled, consented and randomized to the navigator intervention or an informational pamphlet control between 24-34 weeks of gestation. Women randomized to the intervention arm will receive two 20 minute sessions with a trained patient navigator who will guide women in navigating and interpreting information about the quality of care provided at local pediatric practices on the Massachusetts Health Quality Partners web site. A survey designed for the purpose of this study will be administered at baseline and post-intervention. Health literacy, numeracy and level of activation for self-management of health care will also be assessed as potential mediators of intervention effectiveness. The primary study outcome will be the average performance on quality measures for the practices selected in the intervention and control groups. Secondary outcomes will include analyses of efficacy among groups of women defined by parity and an assessment of the relative importance of factors considered when choosing a pediatric care provider. Successful completion of the study aims will yield important new knowledge about the value of guided web-site navigation as a strategy to reduce disparities in the use of publicly reported information.

ELIGIBILITY:
Inclusion Criteria:

* 20-34 weeks of pregnancy
* comfortable speaking English
* ages 16-50

Exclusion Criteria:

* age 15 or younger
* age 51 or greater
* not comfortable speaking or understanding English
* less than 20 or greater than 34 weeks of pregnancy

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 746 (Actual)
Dates: Start 2013-05; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Quality score of pediatric practices chosen by participants | 6-20 weeks
  Each pediatric practice will be given a composite clinical quality and patient experience score based upon scores reported on the Massachusetts Health Quality Partners "Quality Insights" reports. The mean scores of practices chosen by women in the intervention compared to the control arm will assessed.

SECONDARY OUTCOMES:
Factors important to pregnant women when choosing a pediatric practice | 6-20 weeks
  The study survey will assess relative importance of a range of factors that might be important to women when selecting a pediatric practice.

OTHER OUTCOMES:
Patient activation | 6-20 weeks
  We will be assessing changes in patients engagement in self-management of their and their child's health care using Patient Activation Measures.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Goff, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

REFERENCES:
- [Derived] Goff SL, Mazor KM, Guhn-Knight H, Budway YY, Murphy L, White KO, Lagu T, Pekow PS, Priya A, Lindenauer PK. Factors That Matter to Low-Income and Racial/Ethnic Minority Mothers When Choosing a Pediatric Practice: a Mixed Methods Analysis. J Racial Ethn Health Disparities. 2017 Dec;4(6):1051-1060. doi: 10.1007/s40615-016-0309-x. Epub 2017 Mar 8. PMID 28275998
- [Derived] Goff SL, Mazor KM, Pekow PS, White KO, Priya A, Lagu T, Guhn-Knight H, Murphy L, Youssef Budway Y, Lindenauer PK. Patient Navigators and Parent Use of Quality Data: A Randomized Trial. Pediatrics. 2016 Oct;138(4):e20161140. doi: 10.1542/peds.2016-1140. Epub 2016 Sep 6. PMID 27600316
- [Derived] Goff SL, Youssef Y, Pekow PS, White KO, Guhn-Knight H, Lagu T, Mazor KM, Lindenauer PK. Successful Strategies for Practice-Based Recruitment of Racial and Ethnic Minority Pregnant Women in a Randomized Controlled Trial: the IDEAS for a Healthy Baby Study. J Racial Ethn Health Disparities. 2016 Dec;3(4):731-737. doi: 10.1007/s40615-015-0192-x. Epub 2016 Apr 11. PMID 27068662
- [Derived] Goff SL, Pekow PS, White KO, Lagu T, Mazor KM, Lindenauer PK. IDEAS for a healthy baby--reducing disparities in use of publicly reported quality data: study protocol for a randomized controlled trial. Trials. 2013 Aug 7;14:244. doi: 10.1186/1745-6215-14-244. PMID 23919671